CLINICAL TRIAL: NCT03918525
Title: Diabetes In Sindhi Families In Nagpur (DISFIN): An Observational Study
Brief Title: Diabetes In Sindhi Families In Nagpur (DISFIN)
Acronym: DISFIN
Status: Completed | Type: Observational
Sponsor: Lata Medical Research Foundation, Nagpur (Other)
Responsible Party: Sponsor
Other Study IDs: RPC#23A
Record Dates: First submitted 2019-03-13; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 10 ml of venous blood from the ante-cubital vein. This blood sample will be used for lipid profile studies (total and free serum cholesterol, serum triglycerides, high-density lipoproteins, low-density lipoproteins, very low-density lipoproteins and apolipoproteins), fasting plasma glucose, serum cotinine (to corroborate the history of smoking), serum creatinine (to quantify urinary dilution), serum C peptide (to distinguish between type 1 and type 2 diabetes), plasma insulin and serum HbA1c (glycated hemoglobin).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sindhi families — It is an observational study and no intervention is involved

SUMMARY:
The pandemic of diabetes is increasing at an alarming rate. The prevalence of diabetes has risen in India by 123% over the last decade. In 1990, diabetes was not considered an important contributor to mortality in India but in 2013, it is ranked as the eighth most common cause of deaths in adult Indian population. There is now a growing understanding that diabetes runs in families and has a significant genetic basis. In this regard, it is noteworthy that from an ethnographic standpoint, Sindhi population in India has been both genetically and environmentally at an increased risk of stress, hypertension and cardiovascular diseases. Considering the nexus of metabolic diseases that include hypertension, obesity, dyslipidemia and diabetes it is therefore expected that this population may be at an increased risk of these metabolic conditions. However, exact prevalence of contributors to type 2 diabetes in the Sindhi population is unknown. The proposed study will estimate prevalence of type 2 diabetes in Sindhi families of Nagpur. Both the PIs have extensive experience with family studies which includes construction of pedigrees, using variance components methods, dissecting out genetic and environmental components of diseases and association of critical phenotypic traits with disease. The proposed study will tap this resource with a focus on the Sindhi families of Nagpur which are concentrated in the Jaripatka and Khamla areas. This study will exploit the current infrastructure in the Lata Medical Research Foundation to access these families and conduct a first-of-its-kind study in India. It is expected that this study will pave way for more extensive genetic, epigenetic and environmental studies of this population. It will also foster future collaborations with national and international health agencies. In that vein, the DISFIN pilot study represents the first step towards identification, quantification, prevention and control of type 2 diabetes in central India.

DETAILED DESCRIPTION:
At each Participant Recruitment Center:

1. We announced the dates of recruitment locally through pamphlet distribution, personal conversations, emails and a study website to the residents of the study areas. When the participants came in for the study, they were first administered the informed consent form.
2. Upon receiving such consent a Field Research Officer (FRO) appointed specifically for the study collected the demographic data and conduct anthropometric measurements. All the data has been directly input into a cloud-based database through tablet computers made available to the FROs for the purpose of the study.
3. A trained nurse then measured the blood pressure of the participant as follows: These measurements were conducted using a random-zero sphygmomanometer on the left arm. To account for the potential variability in the blood pressure measurements, we measured the blood pressure thrice with 5-minute intervals but use the average of the last two readings as the phenotypic trait value. Appearance of the first Korotkov sound and disappearance of the fifth Korotkov sound was considered as the systolic and diastolic blood pressures, respectively.
4. Thereafter the participant were under electrocardiographic evaluation. The examination was conducted by a trained ECG technician using a portable ECG machine with limb leads, chest leads and augmented leads. The signal recordings were digitized and stored as digital signal files. Novacode software was used to quantitatively measure important phenotypic traits from the ECG signals.
5. The participant then proceeded to measurement of random blood glucose using a glucometer and disposable test strip. The results are shared with the participant as well as entered directly into the cloud-based database.
6. Then the participant were given a urine sample collection cup. The urine sample was used to estimate urine sugar and microalbuminuria.
7. The participant were then given an appointment for fasting blood studies.
8. On the day of the appointment, a trained laboratory technician appointed for the purpose of the study drew 10 ml of venous blood from the ante-cubital vein. This blood sample will be used for lipid profile studies (total and free serum cholesterol, serum triglycerides, high-density lipoproteins, low-density lipoproteins, very low-density lipoproteins and apolipoproteins), fasting plasma glucose, serum cotinine (to corroborate the history of smoking), serum creatinine (to quantify urinary dilution), serum C peptide (to distinguish between type 1 and type 2 diabetes), plasma insulin and serum HbA1c (glycated hemoglobin).
9. To maximize participation for the fasting blood studies, we sent text reminders to participants before the date of appointment. If the participant cannot make it on the day of appointment then we again sent text and/or telephonic reminders to them for a revised appointment date. We did this for a total of three times before the reminders can be stopped.
10. If the participants were diagnosed with any medical condition during the examination then they were duly referred to expert medical help outside of the DISFIN study. If the participant was newly diagnosed as a case of T2D during study the participant was referred to expert diabetologist in the city for further medical care.
11. Lastly, we provided a nominal time compensation for each participant who completed all the study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Resident of Jaripatka or Khamla areas of Nagpur
2. Self-reported Sindhi
3. Age ≥20 years
4. Has given informed consent

Exclusion Criteria:

1. Pregnant or lactating woman
2. Known type 1 diabetes

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To facilitate centralized data and sample collection, we established two Participant Recruitment Centers - one each in Jaripatka and Khamla. These Centers were equipped with facilities to conduct interviews, collect anthropometric data, conduct random blood sugar measurements and collect blood and urine samples for transport and storage.
Sampling Method: Probability Sample
Enrollment: 1462 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Type 2 diabetes | March 1, 2016 - Feb 28, 2017
  Presence of T2D will be defined as: Self-report or FPG ≥126 mg/dl or currently receiving antidiabetic drugs or HbA1c ≥6.5% or random blood sugar ≥ 200 mg/dl

SECONDARY OUTCOMES:
Insulin resistance | March 1, 2016 - Feb 28, 2017
  Insulin resistance will be measured using the Homeostatic Model of Assessment-Insulin resistance (HOMA_IR)
Hypertension | March 1, 2016 - Feb 28, 2017
  Hypertension will be defined using the 2017 revised criteria (systolic blood pressure >120 mmHg and/or diastolic blood pressure >80 mmHg)
Obesity | March 1, 2016 - Feb 28, 2017
  Obesity will be defined as body mass index (BMI) exceeding 30 Kg/m2. BMI will be calculated as weight (in Kg)/Height2 (in meters).
Central obesity | March 1, 2016 - Feb 28, 2017
  Central obesity will be defined using population-specific cut off for waist circumference. For Asian Indians, the cutoffs are: male (>=90cm) and female (>=80 cm).
Dyslipidemia | March 1, 2016 - Feb 28, 2017
  We will use the definition of dyslipidemia as described by the International Diabetes Federation (IDF). The criteria use dyslipidemia is a composite outcomes based on measured values of serum triglycerides (≥ 150 mg/dLmg/dl) and high density lipoprotein (HDL) cholesterol (< 40 mg/dL (1.03 mmol/L) in males < 50 mg/dL (1.29 mmol/L) in females). Additionally, total serum cholesterol (≥200 mg/dl) will also be considered as dyslipidemia.

CONTACTS AND LOCATIONS:
Overall Officials: Manju R Mamtani, MD, Principal Investigator — Treasurer
Locations (1):
- Lata Medical Research Foundation, Nagpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided